CLINICAL TRIAL: NCT01717508
Title: Examination of the Neural Components Underlying the Treatment of Adolescent Major Depression
Brief Title: Neural Components Underlying the Treatment of Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Randy P. Auerbach, Principal Investigator, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012P001844; 2011A053424 (Other Grant/Funding Number: Harvard Medical School); 2011A051965 (Other Grant/Funding Number: McLean Hospital); 2010A054978 (Other Grant/Funding Number: Katz Family Foundation); K23MH097786 (NIH)
Record Dates: First submitted 2012-10-23; First posted 2012-10-30 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Major Depressive Disorder
Keywords: MDD; depression; major depressive disorder; adolescent
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Other): 12 weekly sessions of cognitive behavioral therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Healthy Controls (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 12 sessions of cognitive behavioral therapy
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The goal of the study is to examine how cognitive behavioral therapy (CBT), a common treatment for adolescent depression, affects brain functioning. Depressed adolescents will complete an initial assessment consisting of an interview, questionnaires, computer tasks, and an EEG recording. EEG (electroencephalography) measures brain activity by recording the electrical activity along the scalp caused by the firing of neurons within the brain. They will then complete 12 sessions of cognitive behavioral therapy, which will be 50 minutes long and held once a week for 12 weeks. Before their third therapy session, participants will complete a computer task while EEG data are recorded. After completing the treatment, the participants will complete a final assessment, which will include questionnaires, computer tasks, and an EEG recording. They will also complete follow-up assessments over the phone 1, 3, and 6 months after completing the treatment.

This study will also include healthy control participants. They will complete an initial assessment consisting of an interview, questionnaires, computer tasks, and an EEG recording. Three weeks later, they will return to complete a behavioral task while EEG data are recorded. Twelve weeks after the initial assessment, they will complete a final assessment, which will include questionnaires, computer tasks, and an EEG recording.

DETAILED DESCRIPTION:
The purpose of the study is to examine the impact of individual cognitive behavioral therapy (CBT) for adolescent depression on neural functioning. Specifically, the study will utilize Brent and Poling's (1997) cognitive behavioral therapy (CBT) manual (Cognitive Therapy Treatment Manual for Depressed and Suicidal Youth), and investigators will examine pre- to post- neural activity patterns for children and adolescents who receive individual CBT for depression. Electroencephalography (EEG) techniques will be utilized to assess treatment-related effects on brain activity (i.e., anterior cingulate cortex and dorsolateral prefrontal cortex functioning). Neural activity patterns will also be compared to non-depressed, healthy controls.

ELIGIBILITY:
Inclusion Criteria, Major Depressive Disorder Participants:

* Ages 13-18 years at time of initial assessment
* Female
* Current major depressive disorder (MDD) diagnosed according to the K-SADS Axis I semi-structured interview
* English as first language or English fluency

Exclusion Criteria, Major Depressive Disorder Participants:

* Male
* Mania/Hypomania
* Current anxiety disorders [e.g., Panic Disorder (PD), Generalized Anxiety Disorder (GAD), Obsessive Compulsive Disorder (OCD)]
* Eating Disorders
* Substance Abuse/Dependency
* Conduct Disorder/Antisocial Disorder
* ADHD
* Psychosis
* Mental Retardation
* Organic Brain Syndrome
* Current Psychotherapy Treatment
* Medical & neurological illness (head injury, loss of consciousness for more than 5 minutes, seizures)
* Current use of psychotropic medication for treatment of MDD with the exception of SSRIs (selective serotonin reuptake inhibitors)
* Active suicidality

Inclusion Criteria, Healthy Control Participants:

* Ages 13-18 years at time of initial assessment
* Female
* English as first language or English fluency

Exclusion Criteria, Healthy Control Participants (in addition to the exclusion criteria of the MDD group):

* Elevated depressive symptoms as assessed in phone screen

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2012-10; Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
EEG Activity | 12 weeks
  EEG and ERP measures collected during resting state and behavioral tasks

CONTACTS AND LOCATIONS:
Overall Officials: Randy P Auerbach, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No